CLINICAL TRIAL: NCT05074433
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Anti-Spike SARS-CoV-2 Monoclonal Antibodies as Pre-Exposure Prophylaxis to Prevent COVID-19 in Immunocompromised Participants
Brief Title: A Study to Evaluate Efficacy and Safety of Casirivimab+Imdevimab (Monoclonal Antibodies) for Prevention of COVID-19 in Immunocompromised Adolescents and Adults
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Emerging SARS-CoV2 variants impacting susceptibility to study drug
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: R10933-10987-COV-2176; 2021-005222-14 (EudraCT Number)
Record Dates: First submitted 2021-10-08; First posted 2021-10-12 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Immunocompromised
Keywords: Non-response to COVID-19 vaccination; COVID-19; Immunocompromised, weakened immune system
MeSH Terms: conditions — COVID-19 | interventions — casirivimab and imdevimab drug combination; casirivimab; imdevimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- casirivimab+imdevimab Initial + Q4W (Experimental): Initial subcutaneous (SC) dose, then SC dose every 4 weeks (Q4W)
  Interventions: Drug: casirivimab+imdevimab
- casirivimab+imdevimab Q4W (Experimental): SC dose Q4W
  Interventions: Drug: casirivimab+imdevimab
- casirivimab+imdevimab Q12W (Experimental): SC dose every 12 weeks (Q12W)
  Interventions: Drug: casirivimab+imdevimab
- Placebo (Placebo Comparator): SC dose Q4W
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: casirivimab+imdevimab — Co-administered sequentially subcutaneous (SC)
  Other Names: REGN-COV2; REGN10933; REGN10987; REGEN-COV™; Ronapreve™
  Arms: casirivimab+imdevimab Initial + Q4W; casirivimab+imdevimab Q12W; casirivimab+imdevimab Q4W
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the effect of casirivimab+imdevimab, compared with placebo, in preventing symptomatic SARS-CoV-2 infection in immunocompromised participants.

The secondary objectives of the study are:

* To evaluate the safety and tolerability of repeated SC injections of casirivimab+imdevimab in the study population
* To characterize concentrations of casirivimab and imdevimab in serum over time
* To assess the immunogenicity of casirivimab and imdevimab

ELIGIBILITY:
Key Inclusion Criteria:

1. Meets ≥1 of the following criteria:

   * Is immunocompromised, including people with transplant, who have cancer, primary immunodeficiencies, HIV, rheumatological disease, autoimmune disease, multiple sclerosis OR
   * Currently taking immunosuppressant drugs
2. Have been fully vaccinated against COVID-19 or deemed medically ineligible to receive full course of vaccine
3. Has documented negative serology/antibody response in an anti-SARS-CoV-2 spike protein IgG clinical test or ≤50 U/mL on the Elecsys® SARS-CoV-2 S Total Ig test
4. Tested negative for the COVID-19 virus within 72 hours prior to randomization

Key Exclusion Criteria:

1. Weighs <40 kg (only applies to participants ≥12 to <18 years of age)
2. Has any signs or symptoms consistent with COVID-19
3. Past COVID-19 infection within 90 days prior to randomization
4. Planned use of any investigational, authorized, or approved vaccine for COVID-19 within 90 days of the last dose of study drug
5. Prior, current, or planned use of any of COVID-19 convalescent plasma, other monoclonal antibodies against SARS-CoV-2 or any COVID-19 treatment
6. Is planned to begin immunoglobulin (IVIG) or immunoglobulin (SCIG) therapy, is planned to have a change to existing IVIG or SCIG, or has been on a chronic stable dose of their IVIG or SCIG regimen for less than 90 days prior to screening
7. Has any known active acute respiratory infection
8. Has persistent (refractory to treatment for ≥14 days) bacterial or fungal infection
9. Has known allergy or hypersensitivity to components of the study drugs

NOTE: Other Protocol Defined Inclusion/Exclusion Criteria Apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (67):
- United States (66):
  - Central Alabama Research, Birmingham, Alabama
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Regeneron Study Site, Long Beach, California
  - Regeneron Study Site, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, Sacramento, California
  - Regeneron Study Site, Stanford, California
  - James R Berenson MD Inc., West Hollywood, California
  - University Of Colorado, Aurora, Colorado
  - Regeneron Study Site, North Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Elixia COVID-19, Hollywood, Florida
  - AppleMed Research Group, LLC, Miami, Florida
  - De La Cruz Research Center, LLC, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Florida Medical Clinic, LLC, Zephyrhills, Florida
  - Regeneron Study Site, Atlanta, Georgia
  - Regeneron Study Site, Marietta, Georgia
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Tulane University, New Orleans, Louisiana
  - Institute of Human Virology, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Laboratory of Clinical Immunology and Microbiology, NIAID, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Regeneron Study Site, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Holy Name, Teaneck, New Jersey
  - Maimonides Cancer Center, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Regeneron Study Site, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Regeneron Study Site 2, New York, New York
  - Regeneron Study Site, Rochester, New York
  - Regeneron Study Site, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Burke Primary Care, Morganton, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Regeneron Study Site, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Penn Prevention Clinical Research Site, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Regeneron Study Site, Providence, Rhode Island
  - West Tennessee Research Institute, Jackson, Tennessee
  - PharmaTex Research, LLC, Amarillo, Texas
  - Central Texas Clinical Research, Austin, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Synergy Group Medical,LLC, Houston, Texas
  - Regeneron Study Site, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Regeneron Study Site, Seattle, Washington
  - Swedish Medical Center- First Hill, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
- Regeneron Study Site, Cuauhtémoc, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matching casirivimab+imdevimab - Subcutaneous (SC) dose every 4 weeks (Q4W)
- Casirivimab+Imdevimab Q4W: casirivimab+imdevimab - Subcutaneous (SC) dose every 4 weeks (Q4W)
- Casirivimab+Imdevimab Q12W: casirivimab+imdevimab - Subcutaneous (SC) dose every 12 weeks (Q12W)
Period: Overall Study
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Started | 16 | 17 | 16 | 17
Completed | 7 | 8 | 9 | 11
Not Completed | 9 | 9 | 7 | 6
Not completed — Adverse Event | 0 | 2 | 0 | 1
Not completed — Sponsor Request | 0 | 1 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Subject Decision | 8 | 6 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W | Total
Number analyzed (Participants) | 16 | 17 | 16 | 17 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (14.16) | 60.0 (12.87) | 59.2 (11.67) | 58.2 (13.99) | 59.4 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 11 | 10 | 43
  Male | 4 | 7 | 5 | 7 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 3 | 8
  Not Hispanic or Latino | 14 | 15 | 14 | 14 | 57
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 16 | 16 | 15 | 14 | 61
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Symptomatic (Broad Term), RT-PCR-confirmed SARS-CoV-2 Infection Cases During the EAP
Description: Cumulative incidence of symptomatic (broad term), RT-PCR-confirmed SARS-CoV-2 infection cases during the Efficacy Assessment Period (EAP)
Time Frame: The EAP was defined as the day from first dose of study drug to day 169 +/- 7 days
Measure: Number (95% Confidence Interval); unit: Cumulative Incidence Percentage
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 16 | 17 | 16 | 17
Cumulative Incidence Percentage | 38.1 [5.7 to 72.2] | 14.3 [2.1 to 37.5] | 30.4 [1.3 to 72.0] | 21.4 [2.4 to 53.0]
Statistical Analysis 1: Comparison: Placebo vs Casirivimab+Imdevimab Initial + Q4W; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.563, 95% CI 2-sided [0.093 to 3.393]
Statistical Analysis 2: Comparison: Placebo vs Casirivimab+Imdevimab Q4W; Test type: Superiority; Cox proportional hazard model; Hazard Ratio (HR) = 0.460, 95% CI 2-sided [0.072 to 2.929]
Statistical Analysis 3: Comparison: Placebo vs Casirivimab+Imdevimab Q12W; Test type: Superiority; Cox proportional hazard model; Cox Proportional Hazard = 0.609, 95% CI 2-sided [0.101 to 3.668]

2. Secondary Outcome: Number of Participants With Grade ≥3 Treatment-emergent Adverse Events (TEAEs) During the EAP
Time Frame: The EAP was defined as the day from first dose of study drug to day 169 +/- 7 days
Population: The safety analysis set (SAF) included all participants who received any study drug; it was based on the treatment received (as treated). Determination of "as treated" was based on the actual study drug received. Treatment compliance/administration and all clinical safety variables was analyzed using the SAF.
Measure: Number; unit: Participants
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 16 | 17 | 16 | 17
Participants | 0 | 0 | 0 | 1

3. Secondary Outcome: Number of Participants With Grade ≥3 Treatment-emergent Adverse Events (TEAEs) During the Follow-Up Period
Time Frame: End of EAP to the end of the Follow-Up Period (Day 169 to 205, approximately ~1 months)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 16 | 17 | 16 | 17
Participants | 1 | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With TEAEs Leading to Study Drug Discontinuation During the EAP
Time Frame: The EAP was defined as the day from first dose of study drug to day 169 +/- 7 days
Measure: Number; unit: Participants
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 16 | 17 | 16 | 17
Participants | 0 | 1 | 0 | 1

5. Secondary Outcome: Number of Participants With TEAEs Leading to Study Drug Discontinuation During the Follow-Up Period
Time Frame: End of EAP to the end of the Follow-Up Period (Day 169 to 205, approximately ~1 months)
Measure: Number; unit: Participants
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 16 | 17 | 16 | 17
Participants | 0 | 1 | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs) During the EAP
Time Frame: The EAP was defined as the day from first dose of study drug to day 169 +/- 7 days
Measure: Number; unit: Participants
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 16 | 17 | 16 | 17
Participants | 0 | 0 | 0 | 1

7. Secondary Outcome: Proportion of Participants With Treatment-emergent Serious Adverse Events (SAEs) During the Follow-Up Period
Time Frame: End of EAP to the end of the Follow-Up Period (Day 169 to 205, approximately ~1 months)
Measure: Number; unit: Participants
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 14 | 15 | 15 | 13
Participants | 1 | 1 | 0 | 1

8. Secondary Outcome: Incidence of Adverse Events of Special Interest (AESIs) During the EAP
Time Frame: The EAP was defined as the day from first dose of study drug to day 169 +/- 7 days
Measure: Number; unit: Participants
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 16 | 17 | 16 | 17
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Concentration of Casirivimab Over Time
Time Frame: Up to 28 days postdose for the Q4W groups and 84 days postdose for the Q12 group
Population: The pharmacokinetic analysis set (PKAS) is defined for each analyte separately and includes all treated participants who received any amount of study drug (active or placebo [SAF]), and who had at least 1 non-missing result of respective total analyte following the first dose of study drug or placebo. The PKAS is based on the actual treatment received (as treated) rather than as randomized.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 15 | 15 | 17
mg/L
  0 Days post-dose | 0 (0) | 0 (0) | 0 (0)
  7 Days post-dose: number analyzed (Participants) | 14 | 14 | 15
  7 Days post-dose | 56.9 (18.2) | 15.3 (3.87) | 11.8 (5.01)
  28 Days post-dose: number analyzed (Participants) | 12 | 11 | 13
  28 Days post-dose | 41.7 (13.6) | 10.7 (3.40) | 10.7 (4.68)

10. Secondary Outcome: Concentration of Imdevimab Over Time
Time Frame: Up to 28 days postdose for the Q4W groups and 84 days postdose for the Q12 group
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 15 | 15 | 17
mg/L
  0 Days post-dose | 0 (0) | 0 (0) | 0 (0)
  7 Days post-dose: number analyzed (Participants) | 14 | 14 | 15
  7 Days post-dose | 51.5 (17.5) | 15.2 (5.37) | 11.7 (6.07)
  28 Days post-dose: number analyzed (Participants) | 12 | 11 | 13
  28 Days post-dose | 35.7 (9.45) | 9.16 (3.37) | 9.16 (4.73)

11. Secondary Outcome: Incidence of Anti-drug Antibodies (ADA) Over Time
Time Frame: Up to 28 days postdose for the Q4W groups and 84 days postdose for the Q12 group
Population: The ADA analysis set (AAS) is defined for each study drug separately and includes all treated participants who received any amount of study drug (active or placebo [SAF]) and had at least 1 non-missing ADA result following the first dose of study drug or placebo. The AAS is based on the actual treatment received (as treated) rather than as randomized.
Measure: Number; unit: Participants
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 11 | 12 | 11 | 13
Participants | 11 | 12 | 11 | 13

12. Secondary Outcome: Incidence of Neutralizing Antibodies (NAb) to Each mAb Over Time
Time Frame: Up to 28 days postdose for the Q4W groups and 84 days postdose for the Q12 group
Population: The NAb analysis sets (NAbAS) comprises all treated participants (active or placebo) that were included in the AAS and tested negative at all ADA sampling times or tested positive at 1 or more post dose ADA sampling times and had at least 1 non-missing post dose NAb result (imputed or analysis result). The ADA analysis set (AAS) includes all treated participants who received any amount of study drug and had at least 1 non-missing ADA result following the first dose of study drug or placebo.
Measure: Number; unit: Participants
Arm/Group | Placebo | Casirivimab+Imdevimab Initial + Q4W | Casirivimab+Imdevimab Q4W | Casirivimab+Imdevimab Q12W
Number analyzed (Participants) | 11 | 12 | 11 | 13
Participants | 11 | 12 | 11 | 13

ADVERSE EVENTS:
Time Frame: From first dose to end of follow up (approximately 7 months)
Groups:
- REGN10933+REGN10987 1200mg Loading Dose and 600mg SC Q4W: Co-administered casirivimab+imdevimab combination therapy, 1200 mg (600 mg per mAb) on day 1, then 600 mg (300 mg per mAb) SC Q4W
- REGN10933+REGN10987 300mg SC Q4W: Co-administered casirivimab+imdevimab combination therapy, 300 mg (150 mg per mAb) SC Q4W
- REGN10933+REGN10987 300mg SC Q12W: Co-administered casirivimab+imdevimab combination therapy, 300 mg (150 mg per mAb) SC Q12W
Arm/Group | Placebo | REGN10933+REGN10987 1200mg Loading Dose and 600mg SC Q4W | REGN10933+REGN10987 300mg SC Q4W | REGN10933+REGN10987 300mg SC Q12W
All-Cause Mortality (participants affected / at risk) | 1/16 | 1/17 | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/16 | 1/17 | 0/16 | 2/17
Other Adverse Events (participants affected / at risk) | 7/16 | 5/17 | 10/16 | 8/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | REGN10933+REGN10987 1200mg Loading Dose and 600mg SC Q4W (N=17) | REGN10933+REGN10987 300mg SC Q4W (N=16) | REGN10933+REGN10987 300mg SC Q12W (N=17)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | REGN10933+REGN10987 1200mg Loading Dose and 600mg SC Q4W (N=17) | REGN10933+REGN10987 300mg SC Q4W (N=16) | REGN10933+REGN10987 300mg SC Q12W (N=17)
COVID-19 (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vaginal infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT05074433/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT05074433/SAP_001.pdf